CLINICAL TRIAL: NCT06851819
Title: The Efficacy and Safety of Tislelizumab in Combination with Chemotherapy(etoposide/cisplatin )± Radiotherapy for Extensive-Stage Oligometastatic Small Cell Lung Cancer, a Randomized，Controlled , Phase II Clinical Trial.
Brief Title: Tislelizumab in Combination with Chemotherapy ± Radiotherapy for Extensive-Stage Oligometastatic Small Cell Lung Cancer.
Acronym: TERE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Wenbin SHEN, MD, Hebei Medical University Fourth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024245
Record Dates: First submitted 2025-02-19; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Small Cell Lung Cancer Extensive Stage
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): Chemotherapy and tislelizumab with Concurrent Chest Radiotherapy or Radiotherapy for oligometastases
  Interventions: Radiation: radiotherapy; Drug: immunechemotherapy
- placebo group (Placebo Comparator): Chemotherapy and tislelizumab with no radiotherapy
  Interventions: Drug: immunechemotherapy

INTERVENTIONS:
Radiation: radiotherapy — Palliative radiotherapy for oligometastases can be combined with chemoradiotherapy and immunomaintenance therapy period. The investigator determines the number, timing and regimen of oligometastases according to the location, size, symptoms and patient tolerance of oligometastases
  Arms: experimental group
Drug: immunechemotherapy — Tislelizumab in Combination With Chemotherapy(etoposide/cisplatin )

SUMMARY:
The goal of this clinical trial is to learn the efficacy and safety of tislelizumab in combination with chemotherapy(etoposide/cisplatin ) ± concurrent radiotherapy for extensive-stage oligometastatic small cell lung cancer. 64 Patients with Extensive-Stage Oligometastatic Small Cell Lung Cancer will be randomly divided into the experimental group (tislelizumab combined with chemotherapy and radiotherapy) and the control group (tislelizumab combined with chemotherapy).Researchers will compare treatment efficacy and safety between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 18 years old;
2. Signed written informed consent;
3. Histologically or cytologically confirmed oligometastatic extensive-stage small cell lung cancer (oligometastasis is defined as the number of distant metastatic organs≤ 3, and the number of metastases ≤ 5; The ninth edition of the AJCC/UICC/IASLC TNM Staging Criteria for Lung Cancer (Annex 1), extensive-stage SCLC for any T stage, any N stage, M1a/b/c or T3-4 cannot be included in a tolerable radiotherapy program due to multiple nodules in the lungs or excessive tumor size);
4. chemotherapy must include a combination of cisplatin and etoposide;
5. Expected survival≥ 12 weeks;
6. ECOG score of 0 or 1 (Annex 2);
7. Weight> 40 kg;
8. At least 1 lesion (no prior radiotherapy) according to RECIST 1.1 guidelines, with a maximum diameter of ≥10 mm as accurately measured by computed tomography (CT) or magnetic resonance imaging (MRI) at baseline (except for lymph nodes, which must be ≥15 mm in their short axis); And the lesion is suitable for repeated and accurate measurement.
9. Have not received anti-tumor therapy in the past;
10. Have adequate organ and bone marrow function,
11. Echocardiography: Left ventricular ejection fraction (LVEF) ≥ low limit of normal (50%)
12. Evidence of postmenopausal status in female patients, or negative urine or serum pregnancy test results in premenopausal female patients. A woman is considered menopausal when she stops menstruation for 12 months without an other medical cause.
13. Within 2 weeks (±1 week) prior to enrollment, the following examinations required for staging must be completed: 1) MRI of the head, CT scan of the chest and upper abdomen, ultrasound of superficial lymph nodes and whole-body ECT; Whole-body PET/CT scan is done if necessary.
14. Patients with asymptomatic or stable brain metastases after treatment are allowed to enroll, and patients are required to do not need glucocorticoid therapy or discontinue glucocorticoids within 3 days before the first study dose.

Exclusion Criteria:

1. Personnel involved in the design and/or conduct of this study.
2. Previous receipt of investigational drug in this study.
3. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up phase of an interventional study.
4. There are medical contraindications to etoposide-platinum-based chemotherapy.
5. History of thoracic radiotherapy prior to systemic therapy.
6. Concomitant administration of any chemotherapy, biologics, or hormonal therapy for cancer treatment. Hormone therapy for noncancer-related conditions, such as hormone replacement therapy, is acceptable.
7. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose.
8. History of allogeneic organ transplantation.
9. Patients who have been cured of aplastic anemia or other blood diseases and patients who have undergone stem cell transplantation.
10. Have an autoimmune paraneoplastic syndrome (PNS) that requires systemic therapy (systemic steroids or immunosuppressants) or have clinical symptoms suggestive of an exacerbation of PNS.
11. Active or previously documented autoimmune or inflammatory disease (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [except diverticular disease], systemic lupus erythematosus, Sarcoidosis syndrome, nephrotic syndrome or nephritis, Wegener syndrome [granulomatous vasculitis, Graves' disease, rheumatoid arthritis, hypophysitis and uveitis, etc.]). The following exceptions are made to this criterion: patients with vitiligo or alopecia; Patients with hypothyroidism (e.g., after Hashimoto syndrome) who are stable after receiving hormone replacement therapy; Any chronic skin condition that does not require systemic therapy; Patients with no active disease in the past 3 years may be included in the study after discussion with the study physician; Patients with celiac disease who can be controlled by diet alone.
12. Uncontrolled intercurrent illness including, but not limited to: persistent or active infection, interstitial lung disease, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina, cardiac arrhythmia, severe chronic gastrointestinal disease with diarrhea, or psychiatric/social problems that may limit compliance with study requirements, recent (within 3 months) new cerebral infarction/intracerebral hemorrhage, psychiatric/social problem conditions that result in a significantly increased risk of AEs, or affect the subject's ability to provide written informed consent.
13. History of another primary malignancy, with the following exceptions: malignancy treated with curative intent, no known active disease for 5 years ≥ prior to the first dose and a low risk of potential recurrence; adequately treated non-melanoma skin cancer or lentigo maligna nevus with no evidence of disease; Carcinoma in situ that has been adequately treated and has no evidence of disease.
14. History of leptomeningeal carcinoma.
15. History of active primary immunodeficiency.
16. Active infection, including tuberculosis (clinical evaluation, including clinical history, physical examination, imaging findings, and TB examination consistent with local clinical practice), hepatitis B (known to be HBV surface antigen [HbsAg] positive), hepatitis C, or human immunodeficiency virus (HIV1/2 antibody positive). Patients with prior HBV infection or who have been cured (defined as the presence of hepatitis B core IgG antibodies and the absence of HBsAg) are eligible. Patients who are positive for hepatitis C virus (HCV) antibodies are eligible only if they are negative for HCV RNA polymerase chain reaction.
17. Female patients who are pregnant or lactating.
18. Those who are considered inappropriate by the investigator to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2years
  Progression free survival

SECONDARY OUTCOMES:
Overall survival | 2years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No